CLINICAL TRIAL: NCT04187261
Title: Hip Fractures Surgical Management and Complications: Retrospective Study
Brief Title: Audit of Hip Fractures Surgically Managed
Status: Recruiting | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Obada Hasan, FCPS, MRCS, MSc (Epidemiology&Biostatistics), Primary Investigator, Aga Khan University
Other Study IDs: 4543 21-dec-16
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hip fracture surgeries — fixation or replacement

SUMMARY:
Investigators are reviewing the the charts and medical records of participants who were operated at our institute from 2010 onward for hip fractures. Checking their outcomes (Postoperative complications, length of hospital stay and mortality) and studying their background characteristics and potential associated factors.

DETAILED DESCRIPTION:
This retrospective study is a cohort with multiple exposures and groups. From this nested case control will be analysed as well.

ELIGIBILITY:
Inclusion Criteria:

* All patients, regardless of gender, commodities and age
* Hip fractures which were managed surgically.
* operated at our institute.

Exclusion Criteria:

* Participants with incomplete data or missing information in either the primary exposure or the outcome of interest.
* Participants with pathological fracture, open fractures, poly-trauma or revision surgeries.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: mostly elderly with hi fractures. However we included young patients as well.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 30 days postoperative
  minor or major, in-hospital or within 30 days postoperativel

CONTACTS AND LOCATIONS:
Overall Officials: Obada Hasan, FCPS, MSc, Principal Investigator — Aga Khan Univeristy
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
not allowed by organisation